CLINICAL TRIAL: NCT02599077
Title: Impact vs. Dienogest: A Combined Oral Contraceptive in the Size of Endometriomas in Women With Diameters Smaller Than 4 Centimeters Thereof, at University Hospital Fundación Santa Fe de Bogota, Between the Years 2015-2017
Brief Title: Impact vs. Dienogest: A Combined Oral Contraceptive in the Size of Endometriomas
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fundación Santa Fe de Bogota (Other)
Responsible Party: Principal Investigator, RICARDO RUEDA, gynecologist, Fundación Santa Fe de Bogota
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FSantafeBogota
Record Dates: First submitted 2015-11-03; First posted 2015-11-06 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Endometriosis
Keywords: oral contraceptives; endometrioma; dienogest
MeSH Terms: conditions — Endometriosis | interventions — dienogest; Levonorgestrel; Cyproterone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dienogest (Experimental): the patient handling with 2 mg dienogest / day.
  Interventions: Drug: Dienogest
- Levonorgestrel + ethinylestradiol (Active Comparator): The patient handling with levonorgestrel + ethinylestradiol (0,10 mg - 0,02 )
  Interventions: Drug: Levonorgestrel

INTERVENTIONS:
Drug: Dienogest — patients assigned to this treatment receive 2 milligrams per day
  Other Names: visanne
  Arms: Dienogest
Drug: Levonorgestrel — patients assigned to this treatment receive (0.10 mg levonorgestrel + ethinyl estradiol - 0.02 milligrams daily)
  Other Names: diane
  Arms: Levonorgestrel + ethinylestradiol

SUMMARY:
Project Summary Endometriosis is a disease with a high prevalence that primarily affects women of childbearing age. This condition brings an important physical and emotional burden on sufferers and this is why it requires proper and timely medical management. At present there are several first-line drugs available for the management of symptoms and disease control. In the world literature we have reported several studies that demonstrate the effectiveness of different groups of drugs such as oral contraceptives, progestins, GnRH analogues and danazol. Within the available scientific evidence it has been extensively described the benefits of the new progestins Dienogest, demonstrating a favorable safety profile and efficacy along with a significant reduction of the symptoms of the disease by its anti-inflammatory, and antiproliferative antiagiogénicas in the endometrial tissue . However, although the therapeutic properties of this drug are known, studies are needed to compare its effectiveness with the effectiveness of other therapeutic agents as oral contraceptives. That is why the main objective of this study is to evaluate the impact of Dienogest to 2 mg / day compared with a combined oral contraceptive (levonorgestrel + ethinyl estradiol) in the size of the endometriomas diagnosed by transvaginal ultrasonography in 50 women having diameters less than 4 centimeters of the same, which medical management will be given for one year at the University Hospital Fundación Santa Fe de Bogota. The study was conducted by a clinical trial, randomized, single-blind by the observer. The results will be analyzed and the findings in the study will serve as a tool to define new therapeutic conduct in the management of endometriosis.

DETAILED DESCRIPTION:
Problem and Justification:

Endometriosis is defined as the presence of endometrial tissue outside the uterine cavity, which induces a chronic inflammatory response.

It is a common problem that affects about 6-10% of women of reproductive age, 50-60% of women and adolescents with pelvic pain and nearly 50% of women with infertility. it is characterized by abdominal pain, back pain, pain during sex, dysfunctional uterine bleeding and infertility. Being a common condition among women of childbearing age, which often goes undiagnosed for many years. This delay in diagnosis is due to the variability of symptoms and the lack of tools for accurate diagnosis available for primary care, which is a major burden on the quality of life of patients symptomatic.

The diagnosis of endometriosis should start with clinical history and physical examination and transvaginal ultrasound has proven useful in the diagnosis of ovarian endometriomas and its differential diagnosis with other ovarian masses.

Histologically the lesions identified in endometriosis resemble endometrial tissue in places outside the endometrium, which proliferates in response to hormonal changes that occur with menstruation, causing increased pain and bleeding.

Pharmacological agents are preferred as first-line treatment for managing the symptoms. Among these, oral contraceptives are used to treat symptoms of menorrhagia and dysmenorrhoea associated with endometriosis, affecting the endometrial lining by decreasing the proliferation of endometrial tissue during the menstrual cycle, to shorten the number of days in which endometrial tissue appears, reducing the amount and consistency of bleeding.

Another drug that is used to manage this condition is the Dienogest, which has proven superior to treatment with placebo and the effect is comparable to that of other drugs used in the management of endometriosis, as progestins or GnRH analogues.

All drug treatments for endometriosis are effective in reducing the size and number of lesions, and are not intended to cure the disease or eliminate the injury of the peritoneal cavity. Another management option is surgery, which should be reserved for specific cases or those patients who do not respond to drug treatment.

Endometriosis is a disease that imposes a severe financial burden on society, and a physical and emotional toll on people who have it. Therefore it is important to understand, and education by medical staff against this disease. According to the statistics service approximately 200 women a year are treated in reproductive age of which on average 50 are endometriomas and since there is no clear scientific evidence on the impact of combined oral contraceptives compared with using Dienogest, the objective of this study is to determine the impact of Dienogest to 2 mg / day compared with combined oral contraceptives (levonorgestrel + ethinyl estradiol) in reducing the size of the endometriomas diagnosed by transvaginal ultrasound in women with diameters smaller than 4 centimeters thereof, in the Hospital Universitario Fundación Santa Fe de Bogota.

Goals:

General: Determine the impact of Dienogest to 2 mg / day compared with combined oral contraceptives (levonorgestrel + ethinyl estradiol 0.10 mg - 0.02 mg / day) in the treatment of endometriomas diagnosed by transvaginal ultrasound in women with smaller diameters 4 centimeters thereof, at University Hospital Fundación Santa Fe de Bogota.

Specific:

* Determine Decreasing the size of endometriomas Dienogest using as medical treatment for endometriosis.
* Determine Decreased endometriomas size using a combined oral contraceptive as medical treatment for endometriosis.
* Determine Through ultrasound scanning diagnostic tool as the impact of the reduction in size of endometriomas.
* Compare The effect of the Dienogest vs the combined oral contraceptive in time. Methodology Type of study Experimental study single-blind randomized clinical trial by the observer. Universe Endometriomas of patients with diameters smaller than 4 centimeters diagnosed by transvaginal ultrasound in patients presenting to the Santa Fe de Bogota Foundation between 2015 and 2016.

Sample size

To analyze cases of endometriomas in which medical management vs Dienogest be used with oral contraceptives, the sample size is calculated using the estimated sample size with a comparison of proportions between 2 samples with the following information:

N: 200 Proportion: 1.6%, and the estimated prevalence of endometriosis is 8% and 20% of those with endometriomas.

Confidence level: 95% Z2: 1.96 Alpha error 5% No: 22 Estimated loss: 10%

Sample required:

N1: 25 N2: 25

ELIGIBILITY:
Inclusion Criteria:

Women Of childbearing age (this period), without desire for fertility, without treatment for endometriosis in the past three months, with ultrasound diagnosis of endometrioma (unilateral or bilateral) minor diameter to 4 centimeters. Those who do not go to surgical procedure and who choose or who are instructed to follow a medical management. No contraindications to oral contraceptive use, rating and eligibility criteria of WHO 1 (no restriction can be used in all circumstances) or 2 (the advantages of using the method generally outweigh the risks, usually can be used) . And who they entered the University Hospital Fundación Santa Fe de Bogota.

Exclusion Criteria:

Intercurrent cardiovascular-disease or a history of it (arterial thrombosis or current or previous venous thromboembolism, thrombophilic genetic disease), smoking, obesity, kidney failure, SLE, diagnosed or suspected autoimmune diseases and hypertension.

If you have a history of migraine accompanied by eg visual symptoms, slurred speech or weakness or numbness in any part of the body.

If you have diabetes mellitus with blood vessels. If you have or have had pancreatitis (inflammation of the pancreas) associated with high levels of fatty substances in the blood.

If you have jaundice (yellowing of the skin) or severe liver disease. If you have or have had a cancer that may grow under the influence of sex hormones (eg of the breast or genitals).

If you have or have had a liver tumor, benign or malignant. If you have any unexplained vaginal bleeding. If you are pregnant or think you might be. If you are hypersensitive (allergic) to ethinyl estradiol, levonorgestrel, dienogest or any other part.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
the change from baseline in the size of the endometriomas, as determined by the diagnostic tool ultrasound, subsequent to drug treatment | one year
  The change from baseline in the size of the endometriomas, as determined by the diagnostic tool of ultrasound in a year of contraceptive treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lina restrepo, Study Chair — Fundación Santa Fe de Bogota
Locations (1):
- Fundación Santa Fe de Bogota, Bogota, Cundinamarca, Colombia

REFERENCES:
- [Background] Practice Committee of the American Society for Reproductive Medicine. Endometriosis and infertility: a committee opinion. Fertil Steril. 2012 Sep;98(3):591-8. doi: 10.1016/j.fertnstert.2012.05.031. Epub 2012 Jun 15. PMID 22704630
- [Background] Nnoaham KE, Hummelshoj L, Webster P, d'Hooghe T, de Cicco Nardone F, de Cicco Nardone C, Jenkinson C, Kennedy SH, Zondervan KT; World Endometriosis Research Foundation Global Study of Women's Health consortium. Impact of endometriosis on quality of life and work productivity: a multicenter study across ten countries. Fertil Steril. 2011 Aug;96(2):366-373.e8. doi: 10.1016/j.fertnstert.2011.05.090. Epub 2011 Jun 30. PMID 21718982
- [Background] Eskenazi B, Warner ML. Epidemiology of endometriosis. Obstet Gynecol Clin North Am. 1997 Jun;24(2):235-58. doi: 10.1016/s0889-8545(05)70302-8. PMID 9163765
- [Background] Burney RO, Giudice LC. Pathogenesis and pathophysiology of endometriosis. Fertil Steril. 2012 Sep;98(3):511-9. doi: 10.1016/j.fertnstert.2012.06.029. Epub 2012 Jul 20. PMID 22819144
- [Background] Giudice LC. Clinical practice. Endometriosis. N Engl J Med. 2010 Jun 24;362(25):2389-98. doi: 10.1056/NEJMcp1000274. PMID 20573927
- [Background] Ruan X, Seeger H, Mueck AO. The pharmacology of dienogest. Maturitas. 2012 Apr;71(4):337-44. doi: 10.1016/j.maturitas.2012.01.018. Epub 2012 Feb 24. PMID 22364708
- [Result] Harada T, Momoeda M, Taketani Y, Aso T, Fukunaga M, Hagino H, Terakawa N. Dienogest is as effective as intranasal buserelin acetate for the relief of pain symptoms associated with endometriosis--a randomized, double-blind, multicenter, controlled trial. Fertil Steril. 2009 Mar;91(3):675-81. doi: 10.1016/j.fertnstert.2007.12.080. Epub 2008 Jul 23. PMID 18653184